CLINICAL TRIAL: NCT07116096
Title: Effect of Handgrip Strength on Portal Vein Hemodynamics in Patients With Liver Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Provincial People's Hospital (Other Government)
Collaborators: The First Affiliated Hospital of Shanxi Medical University (Other); The Third People's Hospital of Taiyuan (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MZhao
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Portal pressure measurement group (Experimental)
  Interventions: Device: Jamar Hand Dynamometer, Hand Dynamometer
- Doppler Ultrasound Measurement Group (Experimental)
  Interventions: Device: Jamar Hand Dynamometer, Hand Dynamometer
- Endoscopic Ultrasound Measurement Group (Experimental)
  Interventions: Device: Jamar Hand Dynamometer, Hand Dynamometer

INTERVENTIONS:
Device: Jamar Hand Dynamometer, Hand Dynamometer — Jamar Hand Dynamometer, from Illinois, USA. Maximum handgrip strength was measured three times, with each measurement lasting 3 seconds and a 1-minute interval between tests

SUMMARY:
1. Background Handgrip strength , a core indicator of muscle function, has been confirmed to be significantly associated with the clinical prognosis of patients with liver cirrhosis. However, no studies have explored its correlation with portal venous hemodynamics.
2. Objective The purpose of the study is to examine the effects of Handgrip strength on portal vein and left gastric vein pressure, blood flow velocity and direction in patients with liver cirrhosis, as well as its hemodynamic impact on gastroesophageal varices.
3. Method Study Design: Interventional study. Detection Timing: Hemodynamic indices were measured simultaneously after patients achieved their maximum handgrip strength. Participants were divided into three groups based on the assessment methods. Group 1 (Portal Pressure Measurement Group): Before the placement of TIPS, the pressures of the portal vein and left gastric vein were measured, both before and after the handgrip strength test. Group 2 (Doppler Ultrasound Measurement Group): Measurements of portal flow velocity and direction were taken before and after the handgrip strength test, based on Doppler ultrasound. Group 3 (Endoscopic Ultrasound Measurement Group): Measurements of blood flow volume and direction in esophagogastric varices were conducted before and after the handgrip strength test, based on endoscopic ultrasonography. The inclusion and exclusion criteria were described.
4. Elaboration of the Research Hypothesis 4.1. Core Hypothesis The handgrip strength level in patients with liver cirrhosis is correlated with portal venous system hemodynamic indices. Specifically, enhanced handgrip strength may affect portal hypertension and the hemodynamics of varicose veins by improving systemic muscle function or circulatory status.

4.2. Speculation on potential mechanisms Association between muscle function and circulation: As a representative of systemic muscle function, increased handgrip strength may reflect an increase in cardiac output or changes in splanchnic vascular resistance, thereby influencing portal venous hemodynamics.

Effects on varicose veins: Improved handgrip strength may reduce blood flow velocity or diameter of esophagogastric varices by decreasing splanchnic congestion or regulating local vascular tension, thus lowering the risk of variceal rupture and bleeding.

Role of compensatory mechanisms: Muscle wasting is common in decompensated cirrhosis. Patients with higher handgrip strength may have better compensatory capacity, and the degree of hemodynamic disorder in their portal venous system may be less severe.

Conclusion This study uses a multi-method grouping design to first explore the association between handgrip strength and portal venous hemodynamics in cirrhotic patients. The hypothesis is based on the potential regulatory role of muscle function in the circulatory system, which is expected to provide a new non-invasive indicator for clinical assessment of portal hypertension risk.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years old
* Clinically diagnosed with liver cirrhosis
* Endoscopic observation to determine the presence of esophagogastric varices
* Only eligible for the portal vein pressure measurement group if there are no signs of variceal bleeding for at least 14 days
* Participant or guardian is capable of comprehending the study protocol, willing to participate, and able to provide written informed consent

Exclusion Criteria:

* Severe congestive heart failure, or severe untreated valvular heart disease
* Moderate to severe pulmonary hypertension
* Uncontrolled systemic infection
* Lesions (e.g., cysts) or tumors in the liver parenchyma that preclude TIPS creation
* Overt hepatic encephalopathy
* Unrelieved biliary obstruction
* Child-Pugh score > 13
* MELD score > 18
* INR > 5
* Platelet count < 20 ×109/mm3
* No gastrointestinal bleeding (suitable for the ultrasound examination group and the endoscopic ultrasonography group)
* Participants who had undergone hand or wrist surgery within the previous 3 months or were unable to hold the dynamometer with the testing hand were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
portal pressure | through study completion, an average of 3 minutes
left gastric vein pressure | through study completion, an average of 3 minutes
portal flow velocity | Before the handgrip strength test, and during the maximum handgrip strength phase, measurements were conducted at intervals of 15 seconds, 30 seconds, 45 seconds, and 60 seconds after the release of strength related to the HGS
Portal vein blood flow direction | Before the handgrip strength test, and during the maximum handgrip strength phase, measurements were conducted at intervals of 15 seconds, 30 seconds, 45 seconds, and 60 seconds after the release of strength related to the HGS
Blood flow velocity in esophageal varices | through study completion, an average of 3 minutes
Blood flow direction of esophageal varices | through study completion, an average of 3 minutes
Diameter of esophageal varices | through study completion, an average of 3 minutes
Heart rate | through study completion, an average of 3 minutes
blood pressure | through study completion, an average of 3 minutes

SECONDARY OUTCOMES:
Serum albumin | Baseline
Prothrombin time | Baseline
triglyceride | Baseline
Total cholesterol | Baseline
Fasting blood glucose | Baseline
Serum creatinine | Baseline
Platelet count | Baseline
Serum potassium | Baseline
Serum sodium | Baseline
Serum chloride | Baseline
alanine aminotransferase | Baseline
aspartate aminotransferase | Baseline
Total bilirubin | Baseline
height | Baseline
weight | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
The way of sharing IPD: Sharing and email consultation will begin after December 31, 2026.
  Data collection and Management: Case record forms and electronic data captures.
Supporting Information: Study Protocol
Time Frame: Sharing and email consultation will begin after December 31, 2026.